Principal Investigator: Rocio Pereira, MD

**COMIRB No:** 18-2542 **Version Date:** 3/20/24

**Study Title:** Understanding patient engagement and outcomes in the National Diabetes

**Prevention Program** 

You are being asked to be in this research study as a Lifestyle Coach for the National Diabetes Prevention Program at Denver Health. Your participation in the study involves completing this confidential interview, which should take about 45-60 minutes to complete. There are no costs to you to participate. You will also be asked to participate in two more interviews, one in 6 months and again 6 months after that. This research is being paid for by a grant from the National Institutes of Health.

This study is designed to learn more about what things influence how well people do in the National Diabetes Prevention Program and how to make the program even better in the future. Potential benefits include an improved understanding of how to best help patients reduce their risks for developing type 2 diabetes.

The study has minimal risk, limited to the rare but significant risk of loss of confidentiality. Every effort will be made to protect your privacy and confidentiality. Interview data will be completely confidential, and only used by the study team. To mitigate potential risks, we will only present results in aggregate, and all data will be stored on a secure research server maintained by the University of Colorado Denver. Data collected will be de-identified as quickly as possible and securely transferred to the University of Colorado. To facilitate the interview today, I would like your permission to record the interview, which will be professionally transcribed. During transcription, all names will be removed and a file number will be placed instead as an identifier.

Your participation in this research is voluntary; you have a choice about being in this study. You do not have to be in this study if you do not want to be. You may choose not to answer certain questions if you are uncomfortable. You may choose to withdraw at any time without penalty. Declining participation will not penalize you in any way from your employment. Your participation or non-participation in this study will not be shared with your employer.

If you have questions, you can call the principal investigator, Dr. Rocio Pereira, at 303-602-5049 or email to Rocio.Pereira@dhha.org. If you have questions or concerns about your role and rights as a research participant, would like to obtain information or offer input, or would like to register a complaint about this study, you may contact, anonymously if you wish, the Colorado Multiple Institutional Review Board (COMIRB) at 303-724-1055 or email at COMIRB@ucdenver.edu.

By participating in this interview or the questionnaire, you are agreeing to participate in this research study.